CLINICAL TRIAL: NCT06348706
Title: Effect of Dipeptidyl Peptidase- 4 Inhibitors Supplementation on Non-Alcoholic Steatohepatitis in Adolescents With Type 1 Diabetes Mellitus
Brief Title: Effect of Dipeptidyl Peptidase- 4 Inhibitors on Non-Alcoholic Steatohepatitis and Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Prof. of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ain Shams University25032024
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1; NASH
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Dipeptidyl Peptidase 4; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dipeptidyl peptidase-4 inhibitors supplementation (Active Comparator): Intervention group receiving Dipeptidyl peptidase-4 inhibitors supplementation
  Interventions: Drug: Dipeptidyl peptidase 4 (DPP-4) inhibitor
- Control group (No Intervention): Control group not receiving Dipeptidyl peptidase-4 inhibitors supplementation

INTERVENTIONS:
Drug: Dipeptidyl peptidase 4 (DPP-4) inhibitor — Intervention group received Dipeptidyl peptidase-4 (DPP-4) inhibitors supplementation in a dose of 50 mg with main meal for 6 months.
  Other Names: Dipeptidyl peptidase-4 inhibitors
  Arms: Dipeptidyl peptidase-4 inhibitors supplementation

SUMMARY:
Background: Non-alcoholic steatohepatitis (NASH) is an advanced form of non-alcoholic fatty liver disease (NAFLD) that can precipitate to advanced fibrosis and leads to cardiovascular morbidity and mortality. Many patients with type 1 diabetes mellitus (T1DM) had histological evidence of steatosis and met the histological criteria for NASH. Matrix metalloproteinase-14 (MMP-14) is a type 1 transmembrane proteinase expressed in liver fibrosis and is involved in the development of atherosclerosis and cardiovascular disease. Hepatic dipeptidyl peptidase-4 (DPP-4) expression in NAFLD may be directly associated with hepatic lipogenesis and liver injury. Some studies showed the beneficial effect of dipeptidyl peptidase-4 (DDP-4) inhibitors in NAFLD/NASH for their role in improving hepatic glucose metabolism. Vildagliptin, a DPP-4 inhibitor, could be promising therapeutic agents for NAFLD/NASH.

To the best of our knowledge, no previous study assessed the role of DPP-4 inhibitors in adolescent patients with T1DM and NASH.

Objectives: This randomized-controlled clinical trial assessed the impact of the oral DPP-4 inhibitor, vildagliptin, as an add-on therapy on NASH in adolescents with T1DM as well as its effect on glycemic control, lipid profile, MMP-14 levels and CIMT as a marker for subclinical atherosclerosis.

Methods: This study included 60 adolescents with T1DM and NASH with a mean age 15.6 ± 2.08 years and disease duration ≥ 5 years. Forty age- and sex-matched healthy subjects with a mean age 14.9 ± 3.2 years were enrolled as healthy controls to compare MMP-14 levels. T1DM patients were randomly assigned to receive oral vildagliptin (50 mg daily) with lunch meal for six months or not. Fasting and 2 hours post-prandial blood glucose levels, HbA1c, liver function tests, fasting lipid profile, hepatic steatosis index and triglyceride glucose (TyG) index were assessed. MMP-14 levels were measured by enzyme-linked immunosorbent assay among all patients and healthy controls. CIMT was assessed using Doppler ultrasound and transient elastography with controlled attenuation parameter (CAP) was performed to assess liver stiffness and steatosis stage.

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) is characterised by excessive hepatic fat accumulation (steatosis) in the absence of significant alcohol consumption, occurring with or without hepatic inflammation and fibrosis. Steatosis may progress to a more advanced form of the disease, non-alcoholic steatohepatitis (NASH), which can precipitate to advanced fibrosis, leading to cirrhosis and/or hepatocellular carcinoma (HCC) and can result in the need for liver transplantation or death as well as cardiovascular morbidity and mortality.

It was demonstrated that 53.1% of patients with type 1 diabetes mellitus (T1DM) had histological evidence of steatosis and 20.4% met the histological criteria for NASH. Patients with T1DM onset at an earlier age have an increased incidence of cardiovascular disease (CVD) events and increased CVD mortality.

Matrix metalloproteinases (MMPs) are found to have multiple biological activities including diseases like angiogenesis and cirrhosis. They are expressed in atherosclerotic plaques, promoting vascular remodelling, contributing to atherothrombosis, and plaque disruption. MMP-14 is involved in the development of atherosclerosis and CVD. MMP-14 is also noticed to be expressed in highly invasive hepatocellular carcinoma and expressed in liver fibrosis.

Carotid ultrasound is easily available, a cost effective and non-invasive tool for evaluating carotid artery intima-media thickness (CIMT) to assess CVD as carotid atherosclerosis. CIMT was higher for individuals with NASH than for those with simple steatosis.

Dipeptidyl peptidase-4 (DPP-4) inhibitors are a relatively new class of oral diabetes drugs with a glucose-lowering effect. DPP-4 inhibitors exert their glucose-lowering effects primarily by blocking the enzyme DPP-4, which is involved in the degradation of incretins, including glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP). DPP-4 inhibitors are widely used for the treatment of type 2 diabetes since 2006. Although DPP-4 inhibitors may be beneficial for T1DM, existing studies do not strongly support these positive effects in clinical practice.

Vildagliptin, an oral antihyperglycemic agent that competitively inhibits DPP-4. A few trials have demonstrated that vildagliptin has an effect on NAFLD. In 44 patients with T2DM and hepatic steatosis, vildagliptin treatment for 6 months decreased liver enzymes and intrahepatic triglyceride content, as assessed by MRI. In a study conducted in Pakistan, vildagliptin for 12 weeks improved liver enzymes and steatosis grading, as assessed by ultrasound.

Aim: To assess the effect of Dipeptidyl peptidase-4 (DPP-4) inhibitors supplementation as an add on therapy on NASH in adolescents with type 1 diabetes mellitus as well as its effect on glycemic control, lipid profile, MMP-14 levels and CIMT as a marker for subclinical atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents diagnosed with type 1 diabetes according to ISPAD guidelines .
* Patients aged 12-18 years with NASH.
* Patients on regular visit to clinic.
* Patients on regular insulin therapy.

Exclusion Criteria:

* Patients with renal impairment due to cause other than diabetes.
* Patients with hypertension.
* Hyper- or hypo-thyroidism.
* Hepatitis virus infection (B or C) or any evidence of infection.
* History of liver disease other than NASH such as cholestasis and Wilson disease.
* Patients with autoimmune hepatitis.
* Recurrent diabetic ketoacidosis (more than 2 episodes in the previous 12 months)
* Patients were already on anti-hypertensive drugs or any antioxidant therapy such as vitamin supplements.
* Taking any vitamins or food supplements one month before study.
* Participation in a previous investigational drug study within 3 months preceding screening.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related effect on NASH status in adolescents with type 1 diabetes mellitus | 6 months
  Effect of DPP-4 inhibitors on NASH in adolescents with type 1 diabetes mellitus measured by Doppler ultrasound and transient elastography with controlled attenuation parameter (CAP) to assess liver stiffness and steatosis stage.

SECONDARY OUTCOMES:
Number of participants with treatment-related Matrix metalloproteinase-14 (MMP-14) level change | 6 months
  Effect of (DPP-4) inhibitors supplementation on Matrix metalloproteinase-14 (MMP-14, (ng/mL) level
Number of participants with treatment-related Glycemic control (HbA1c%) level change | 6 months
  Effect of Dipeptidyl peptidase-4 (DPP-4) inhibitors on glycemic control (HbA1c%)

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Elbarbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Temple JL, Cordero P, Li J, Nguyen V, Oben JA. A Guide to Non-Alcoholic Fatty Liver Disease in Childhood and Adolescence. Int J Mol Sci. 2016 Jun 15;17(6):947. doi: 10.3390/ijms17060947. PMID 27314342
- [Result] Verges B. Cardiovascular disease in type 1 diabetes: A review of epidemiological data and underlying mechanisms. Diabetes Metab. 2020 Nov;46(6):442-449. doi: 10.1016/j.diabet.2020.09.001. Epub 2020 Sep 28. PMID 32998054
- [Result] Geervliet E, Moreno S, Baiamonte L, Booijink R, Boye S, Wang P, Voit B, Lederer A, Appelhans D, Bansal R. Matrix metalloproteinase-1 decorated polymersomes, a surface-active extracellular matrix therapeutic, potentiates collagen degradation and attenuates early liver fibrosis. J Control Release. 2021 Apr 10;332:594-607. doi: 10.1016/j.jconrel.2021.03.016. Epub 2021 Mar 15. PMID 33737203
- [Result] Targher G, Bertolini L, Padovani R, Rodella S, Zoppini G, Zenari L, Cigolini M, Falezza G, Arcaro G. Relations between carotid artery wall thickness and liver histology in subjects with nonalcoholic fatty liver disease. Diabetes Care. 2006 Jun;29(6):1325-30. doi: 10.2337/dc06-0135. PMID 16732016
- [Result] Sumida Y, Yoneda M, Tokushige K, Kawanaka M, Fujii H, Yoneda M, Imajo K, Takahashi H, Eguchi Y, Ono M, Nozaki Y, Hyogo H, Koseki M, Yoshida Y, Kawaguchi T, Kamada Y, Okanoue T, Nakajima A, Jsg-Nafld JSGON. Antidiabetic Therapy in the Treatment of Nonalcoholic Steatohepatitis. Int J Mol Sci. 2020 Mar 11;21(6):1907. doi: 10.3390/ijms21061907. PMID 32168769
- [Result] Wang Q, Long M, Qu H, Shen R, Zhang R, Xu J, Xiong X, Wang H, Zheng H. DPP-4 Inhibitors as Treatments for Type 1 Diabetes Mellitus: A Systematic Review and Meta-Analysis. J Diabetes Res. 2018 Jan 8;2018:5308582. doi: 10.1155/2018/5308582. eCollection 2018. PMID 29507862
- [Result] Hussain M, Majeed Babar MZ, Hussain MS, Akhtar L. Vildagliptin ameliorates biochemical, metabolic and fatty changes associated with non alcoholic fatty liver disease. Pak J Med Sci. 2016 Nov-Dec;32(6):1396-1401. doi: 10.12669/pjms.326.11133. PMID 28083033